CLINICAL TRIAL: NCT02821078
Title: Evaluation of 4D Magnetic Resonance Flow Sequence at Hepatic Level
Acronym: HEPAFLUX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PI2016_843_0010; 2016-A00641-50 (Other: IDRCB)
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Magnetic Resonance Imaging
Keywords: phase-contrast MRI; blood flow; velocity mapping; abdominal imaging; Quantitative MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): In addition to the standard clinical MR protocol, 2 added sequences:
  * 4D flow imaging sequence
  * standard 2D-PhaseContrast at portal trunk level as reference
  Interventions: Other: 4D flow imaging sequence

INTERVENTIONS:
Other: 4D flow imaging sequence — 4D flow imaging sequence

SUMMARY:
The objective of the project is to establish the 3D velocity mapping of the hepatic vasculature and its consistency

DETAILED DESCRIPTION:
The objective of the project is to establish the 3D velocity mapping of the hepatic vasculature and its consistency. Specifically, the investigators will assess the consistency of the quantitative data by measuring hepatic blood Inflow (hepatic artery + portal vein) and outflow (inferior vena cava differential flow). According to the mass conservation physical property, blood inflow must equals blood outflow. The relative gap between the measured values will characterize the consistency of the acquisition.

ELIGIBILITY:
Inclusion Criteria:

* Participants have fasted for 6 hours before examination
* Adult participants

Exclusion Criteria:

* Anyone with a classic contraindication to MRI
* Recanalized umbilical vein
* Severe obesity
* Gadolinium chelate allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Hepatic blood flow difference | Day 0
  difference between (hepatic artery + portal vein flows) and inferior vena cava differential flow (infra and supra hepatic)

SECONDARY OUTCOMES:
Comparison between 4D and 2D flow | Day 0
  Comparison between 4D and 2D flow values measured at the portal trunk level

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Yzet, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yzet T, Bouzerar R, Baledent O, Renard C, Lumbala DM, Nguyen-Khac E, Regimbeau JM, Deramond H, Meyer ME. Dynamic measurements of total hepatic blood flow with Phase Contrast MRI. Eur J Radiol. 2010 Jan;73(1):119-24. doi: 10.1016/j.ejrad.2008.09.032. Epub 2008 Nov 12. PMID 19008062